CLINICAL TRIAL: NCT05255484
Title: A Phase I/II, Open-Label, Dose Escalation and Expansion Study of LM-108 as a Single Agent or in Combination With Pembrolizumab in Advanced Solid Tumors
Brief Title: Study of LM-108 as a Single Agent or in Combination With Pembrolizumab in Subjects With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Completed primary objective.
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM108-01-102
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LM-108 Dose Escalation (Experimental): Drug: LM-108 Administered intravenously
  Interventions: Drug: LM-108
- LM-108 Dose Expansion (Experimental): Drug: LM-108 Administered intravenously
  Interventions: Drug: LM-108
- LM-108 Combination Dose Escalation (Experimental): Drug: LM-108 Administered intravenously Drug: An Anti-PD-1 Antibody Administered intravenously
  Interventions: Drug: LM-108; Drug: An Anti-PD-1 Antibody
- LM-108 Combination Dose Expansion (Experimental): Drug: LM-108 Administered intravenously Drug: An Anti-PD-1 Antibody Administered intravenously
  Interventions: Drug: LM-108; Drug: An Anti-PD-1 Antibody

INTERVENTIONS:
Drug: LM-108 — Administered intravenously
Drug: An Anti-PD-1 Antibody — Administered intravenously
  Arms: LM-108 Combination Dose Escalation; LM-108 Combination Dose Expansion

SUMMARY:
A Phase I/II, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LM-108 as a Single Agent or in Combination with Pembrolizumab in Advanced Solid Tumors

DETAILED DESCRIPTION:
A Phase I/II, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LM-108 as a Single Agent or in Combination with Pembrolizumab in Advanced Solid Tumors

The study schedule includes screening visit (28 days prior to accept the investigational medicinal product (IMP)), treatment visit (accept IMP for the first time to the end of treatment (EOT)/early withdrawal), and follow-up visit (28 days after the EOT/early withdrawal).

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
2. Histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
3. At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
4. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose

Key Exclusion Criteria:

1. Any adverse event from prior anti-tumour therapy has not yet recovered to ≤grade 1 of CTCAE v5.0
2. Uncontrolled tumour-related pain
3. Known central nervous system (CNS)
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
5. Use of inhaled corticosteroids
6. Known history of autoimmune disease
7. Use of any live attenuated vaccines within 28 days
8. Have severe cardiovascular disease
9. Uncontrolled or severe illness
10. History of immunodeficiency disease
11. Active malignancies which are likely to require the treatment.
12. Child-bearing potential female
13. Have psychiatric illness or disorders

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
AEs | 126 weeks
  Incidence of adverse events
DLT | 21 days
  Incidence of dose-limiting toxicity (DLT)
SAE | 126 weeks
  Incidence of serious adverse event
Incidence of clinical significant in laboratory examinations | 126 weeks
  Incidence of clinical significant in laboratory examinations, including hematology, urinalysis, blood biochemistry, coagulation tests and thyroid function.

SECONDARY OUTCOMES:
Incidence of anti-drug antibodies to LM-108 | 126 weeks
  Incidence of anti-drug antibodies to LM-108
Cmax | 126 weeks
  Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) for LM-108
Cmin | 126 weeks
  PK Parameter: Minimum Observed Concentration (Cmin) for LM-108
Tmax | 126 weeks
  PK Parameter: Time of Maximum Observed Concentration (Tmax) for LM-108
AUC | 126 weeks
  PK Parameter: Area Under the Concentration-time Curve (AUC) for LM-108
Cmax,ss | 126 weeks
  PK Parameter: Steady State Maximum Concentration (Cmax,ss)
Cmin, ss | 126 weeks
  PK Parameter: Steady State Minimum Concentration (Cmin, ss)
CLss | 126 weeks
  PK Parameter: Systemic Clearance at Steady State (CLss)
Rac | 126 weeks
  PK Parameter: Accumulation Ratio (Rac)
t 1/2 | 126 weeks
  PK Parameter: Elimination Half-life (t 1/2)
Vss | 126 weeks
  PK Parameter: Volume of Distribution at Steady-State (Vss)
DF | 126 weeks
  PK Parameter: Degree of Fluctuation (DF)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ocala Oncology Center, Ocala, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Gabrail Cancer and Research Center, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Oklahoma, Norman, Oklahoma
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No